CLINICAL TRIAL: NCT05358574
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Anatomical Shoulderᵀᴹ Bipolar System (Implants and Instrumentation) - A Retrospective and Prospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the Anatomical Shoulder Bipolar System
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-130E
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Revision of a Shoulder Prosthesis
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the Anatomical Shoulder Bipolar: Patients who received the Anatomical Shoulder Bipolar and were operated according to the product's IFU and surgical technique

SUMMARY:
The study is a monocentric, retrospective and prospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to collect long-term data confirming safety, performance and clinical benefits of the Anatomical Shoulder Bipolar System (Implants and Instrumentation) when used as a salvage solution in shoulder replacement.

The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcome measures (PROMs) as well as radiographic outcomes.

DETAILED DESCRIPTION:
The Anatomical Shoulder Bipolar System is intended for hemi shoulder replacement as a salvage solution in situations, where a Zimmer Anatomical Shoulder Inverse/Reverse prosthesis was originally planned, but it is intra-operatively found that the attachment of the Zimmer Anatomical Shoulder Inverse/Reverse glenoid fixation is not possible. The system is intended for long-term implantation into the human shoulder joint.

One site will be involved in this study. The aim is to include a maximum of 40 consecutive series cases who received the Anatomical Shoulder Bipolar starting from 2009 until 2020. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop and immediate post-op intervalls will be available in medical notes and collected retrospectively. During follow-up visits at 1, 2, 5, 7 and 10 years post-op (depending on patients' date of surgery), the patient will be asked to complete patient questionnaires. Moreover, a clinical assessment and a radiographic evaluation will be conducted. In addition, any complications and adverse events will also be collected during these follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. The Anatomical Should Bipolar Adaptor is indicated for hemi shoulder replacement as a salvage solution in situations, where a Zimmer Anatomical Shoulder Inverse/Reverse prosthesis was originally planned, but it is intra-operatively found that the attachment of the Zimmer Anatomical Shoulder Inverse/Reverse glenoid fixation is not possible
2. Patient should have received the Anatomical Shoulder Bipolar System
3. Patient should have signed the Informed Consent Form
4. Patient is 18-100 years of age, inclusive
5. Patient is skeletally mature

Exclusion Criteria:

1. Patients who are not willing to return for study required follow-up visits and/or are not willing to comply with the follow-up schedule
2. Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is a known drug abuser, a known alcoholic or anyone who cannot understand what is required of them
3. Patient is known to be pregnant or breastfeeding
4. Musculoskeletal situation that enables the application of a regular hemi or total shoulder system
5. Good quantity or quality of the glenoid bone, where the fixation of a Zimmer Anatomical Shoulder Inverse/Reverse glenoid fixation is possible
6. Patient's physical conditions that would impair achieving adequate implant support, and/or prevent the use of an appropriately sized implant (e.g. due to insufficient quality or quantity of bone).
7. Signs of infection
8. Non-functional deltoid muscle
9. Charcot's shoulder (neuroarthropathy)
10. Presence of significant injury to the upper brachial plexus
11. Any neuromuscular or vascular disease compromising the affected limb that would endanger the success of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of a consecutive series of cases implanted with the Anatomical Shoulder Bipolar System according to Zimmer Biomet's Instruction for Use (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2033-07-16 (Estimated); Study Completion 2033-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and frequency of revisions [Product safety based on implant survivorship] | From operation to study completion, 1-10 years
  Safety will be assessed by recording and analyzing the incidence and frequency of revisions, complications and adverse events. A Kaplan Meier survival curve will be calculated.

SECONDARY OUTCOMES:
Constant and Murley Score | From post-operative to final follow-up visit, 1-10 years
  The patient will be evaluated at each interval (1, 2, 5, 7, 10 years) The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points.
Oxford Shoulder Score | From post-operative to final follow-up visit, 1-10 years
  The patient will be evaluated at each interval (1, 2, 5, 7, 10 years) The OSS is a self-assessment of shoulder pain and function with 12 items; pain (2), interference with pain (2), and daily functions (8). Each response is answered with a five point Likert scale. The total score is the sum of the 12 items, with lower scores indicating a more favorable outcome.
EuroQol Five Dimensions Questionnaire | From post-operative to final follow-up visit, 1-10 years
  The patient will be evaluated at each interval (1, 2, 5, 7, 10 years)
  The EQ-5D measures 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a total of 5 questions. It is accompanied by the patient's self-assessment with the VAS.
  Each dimension is assigned one of three discrete levels for evaluation on the day of administration:
  Level 1 - No problems, no disability Level 2 - Some problems, moderate disability Level 3 - A lot of problems, severe disability
  The final score is a five digit composite of the responses ranging between 33333 - 11111 with 243 possible combinations in between.
X-rays | From post-operative to final follow-up visit, 1-10 years
  Performance and clinical benefits will be assessed by radiographic evaluation. Radiographs (A/P and axillary view) of the operated shoulder will be taken at each interval.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Helios ENDO-Klinik, Hamburg, Germany